CLINICAL TRIAL: NCT02324725
Title: Biomarkers of Disease and Response to Treatment in Opioid Addiction
Brief Title: Biomarkers of Injectable Extended Release Naltrexone Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 814234
Record Dates: First submitted 2014-12-08; First posted 2014-12-24 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Heroin Dependence; Opioid Dependence
Keywords: naltrexone; neuroimaging; heroin; addiction; dependence; opioid; Vivitrol®; functional magnetic resonance imaging
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Behavior, Addictive | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naltrexone Intervention (Experimental): Eligible participants receive up to three monthly injections of 380 mg of naltrexone contained in dissolvable polymer microspheres and administered by deep intramuscular injection and slowly released over a period of approximately 4 weeks.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Up to three monthly injections of 380 mg of naltrexone suspended in dissolvable polymer microspheres and administered intramuscularly
  Other Names: Vivitrol ®

SUMMARY:
This study evaluates the biological markers of treatment of opioid dependent individuals with an extended release formulation of the opioid antagonist naltrexone. The biological measures include functional MRI, blood levels of naltrexone and its metabolites, urine toxicology and behavioral tests probing various aspects of personality, memory, reward processing and attention.

DETAILED DESCRIPTION:
This study is using blood oxygenation level dependent (BOLD) functional magnetic resonance imaging (fMRI) to examine the brain predictors of adherence and outcomes of opioid antagonist therapy. Opioid-dependent intravenous heroin users are offered up to 3 monthly injections of the extended-release naltrexone (XRNTX) contingent upon successful outpatient non-opioid detoxification, with an additional 4 weeks of follow up. Brain responses to heroin-related pictures are recorded using fMRI prior to the 1st XRNTX injection and approximately 2 weeks thereafter the 1st XRNTX injection. Primary clinical variables include the number of injections (maximum of 3) accepted by participants, change in self-reported craving for opioids after exposure to drug-related visual cues during the brain fMRI sessions, urine levels of ten commonly abused substances and self-report of cigarette use.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR diagnosis of opioid dependence, active opioid use, confirmed by urine toxicology screen and self-reported monthly intravenous heroin use for more than 2 weeks in the past 3 months
2. urine toxicology screen negative for opioids after detoxification
3. good physical health as indicated by history and physical examination, screening blood work-up and urinalysis.

Exclusion Criteria:

1. chronic medical illnesses;
2. current use of medications potentially confounding brain activity, such as anti-dopaminergic agents, anti-depressants and beta-blockers;
3. current DSM-IV-TR Axis I psychiatric disorders other than opioid and nicotine dependence;
4. life time history of concurrent IV cocaine and heroin (speedball) administration;
5. pregnancy or breastfeeding;
6. history of clinically significant head trauma;
7. contraindications for naltrexone treatment including medical conditions requiring opioid analgesics, e.g. chronic pain or planned surgery, obesity, elevated liver enzymes (> 3 times upper limit of normal), failure to complete opioid detoxification
8. contraindications for MRI, i.e. indwelling magnetically active foreign bodies and phobia to enclosed spaces

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Brain response to heroin-related visual cues | 1 hour
  Brain, behavioral and motivational (e.g. craving) response to audiovisual drug-related and control stimuli (images, smells and sounds) and to standard tasks of decision making, self-appraisal, response inhibition, social interaction and reward processing.

SECONDARY OUTCOMES:
Cigarettes smoked per day | 6 months
  behavioral
Urine toxicology | 6 months
  Urine toxicology for methamphetamine, amphetamines, cannabis, cocaine, oxycodone, buprenophine, methadone, opioids, benzodiazepines and barbiturates.
Injections | 3 months
  Number of injections (maximum of 3) accepted by participants
Motivational response to opioid-related visual cues measured by self-reported craving for opioids | 2 hours
  Change in self-reported craving for opioids after exposure to opioid-related visual cues during functional MRI sessions

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Langleben, MD, Principal Investigator — Co-Investigator
Locations (1):
- Center for the Studies of Addiction, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang AL, Shi Z, Elman I, Langleben DD. Reduced cigarette smoking during injectable extended-release naltrexone treatment for opioid use disorder. Am J Drug Alcohol Abuse. 2020 Jul 3;46(4):472-477. doi: 10.1080/00952990.2020.1741001. Epub 2020 May 7. PMID 32379516